CLINICAL TRIAL: NCT00605865
Title: Drug Use Investigation of Jzoloft.
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0501090
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Panic Disorder; Depression
MeSH Terms: conditions — Panic Disorder; Depression | interventions — Sertraline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sertraline hydrochloride.: Patients taking Sertraline hydrochloride.
  Interventions: Drug: Sertraline hydrochloride

INTERVENTIONS:
Drug: Sertraline hydrochloride — J ZOLOFT® Tablets 25 mg and J ZOLOFT® Tablets 50 mg. J ZOLOFT is Brand name in Japan.
  Dosage, Frequency: According to Japanese LPD, "The usual initial dose of J ZOLOFT in adults is 25 mg daily as sertraline and then gradually increased up to 100 mg, which should be given orally once daily. The dose may be adjusted within the range not exceeding 100mg according to the patient's age and symptoms".
  Duration: According to the protocol of A0501090, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 16 weeks after the first administration.
  Other Names: J Zoloft, Zoloft

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reactions not expected from the LPD (unknown adverse drug reactions), 2) the incidence of adverse drug reactions in this surveillance, and 3) factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Sertraline hydrochloride should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be taking Sertraline hydrochloride in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not taking Sertraline hydrochloride.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients to whom an investigator involved in A0501090 prescribes sertraline hydrochloride.
Sampling Method: Probability Sample
Enrollment: 2272 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501090&StudyName=Drug%20Use%20Investigation%20of%20Jzoloft.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline: Participants taking Sertraline according to Japanese Package Insert
Period: Overall Study
Arm/Group | Sertraline
Started | 2272
Completed | 2157
Not Completed | 115
Not completed — Protocol Violation | 115

BASELINE CHARACTERISTICS:
Arm/Group | Sertraline
Number analyzed (Participants) | 2157
Age, Customized [Number; unit: participants]
  <65 years | 1820
  >=65 years | 337
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1289
  Male | 868
Target Disease [Number; unit: participants] — The target disease which was diagnosed by investigator
  participants
    Depression/Depressed State | 1870
    Panic Disorder | 150
    Depression/Depressed state and Panic Disorder | 56
    Other than Those Above | 81
Target Disease Severity [Number; unit: participants] — The severity of target disease which was diagnosed by investigator
  participants
    Mild | 568
    Moderate | 1423
    Severe | 166
Complications [Number; unit: participants] — Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
  participants
    Present | 777
    Absent | 1380
Concomitant Drug [Number; unit: participants] — Concomitant drugs is the drugs which participant had taken during the observation period of this study to treat for participant's illnesses, injuries etc. The physician of this survey listed all of concomitant drugs. (e.g. paroxetine, milnacipran, etc.)
  participants
    Present | 1874
    Absent | 283
Starting Dose [Number; unit: participants] — Starting dose of each participant enrolled in this study
  participants
    25 mg | 1530
    50 mg | 523
    75 mg | 33
    100 mg | 31
    Other than Those Above | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants of Treatment Related Adverse Events (TRAEs)
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Time Frame: Baseline up to 16 weeks
Population: Safety analysis population included all enrolled participants who had received at least 1 confirmed administration of Sertraline.
Measure: Number; unit: participants
Groups:
- Sertraline: Participants who took Sertraline according to Japanese Package Insert
Arm/Group | Sertraline
Number analyzed (Participants) | 2157
participants | 263

2. Primary Outcome: Number of Treatment Related Adverse Events (TRAEs) Not Expected From Japanese Package Insert
Time Frame: Baseline up to 16 weeks
Population: The safety analysis population consists of the cases that satisfy the participant's conditions and in whom administration of Sertraline was confirmed.
Measure: Number; unit: events
Arm/Group | Sertraline
Number analyzed (Participants) | 2157
events
  Dyspnoea | 3
  Gastritis | 3
  Sedation | 2
  Erectile dysfunction | 2

3. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Complications
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without complications is significant risk factor, Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Complications: Participants with complications who took Sertraline according to Japanese Package Insert
- Without Complications: Participants without complications who took Sertraline according to Japanese Package Insert
Arm/Group | With Complications | Without Complications
Number analyzed (Participants) | 777 | 1380
participants | 129 | 134
Statistical Analysis 1: Comparison: With Complications vs Without Complications; The risk factor tested was "complications". The null hypothesis is there is no difference between "with and without complications" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

4. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Concomitant Drug
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without concomitant drug is significant risk factor, Concomitant drugs is the drugs which participant had taken during the observation period of this study to treat for participant's illnesses, injuries etc. The physician of this survey listed all of concomitant drugs. (e.g. paroxetine, milnacipran, etc.)
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Concomitant Drug: Participants with concomitant drug who took Sertraline according to Japanese Package Insert
- Without Concomitant Drug: Participants without concomitant drug who took Sertraline according to Japanese Package Insert
Arm/Group | With Concomitant Drug | Without Concomitant Drug
Number analyzed (Participants) | 1864 | 293
participants | 238 | 25
Statistical Analysis 1: Comparison: With Concomitant Drug vs Without Concomitant Drug; The risk factor tested was "concomitant drug". The null hypothesis is there is no difference between "with and without concomitant drug" in the participants of responders; Test type: Superiority or Other; p = 0.039, Chi-squared — not adjusted, p=0.050

5. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Renal Dysfunction
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without renal dysfunction is significant risk factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Renal Dysfunction: Participants with renal dysfunction who took Sertraline according to Japanese Package Insert
- Without Renal Dysfunction: Participants without renal dysfunction who took Sertraline according to Japanese Package Insert
Arm/Group | With Renal Dysfunction | Without Renal Dysfunction
Number analyzed (Participants) | 24 | 2133
participants | 7 | 256
Statistical Analysis 1: Comparison: With Renal Dysfunction vs Without Renal Dysfunction; The risk factor tested was "renal dysfunction". The null hypothesis is there is no difference between "with and without renal dysfunction" in the participants of responders; Test type: Superiority or Other; p = 0.011, Chi-squared — not adjusted, p=0.050

6. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Past Medical History of Other Illness
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without Past Medical History of Other Illness is significant risk factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Past Medical History of Other Illness: Participants with past medical history of other illness who took Sertraline according to Japanese Package Insert
- Without Past Medical History of Other Illness: Participants without past medical history of other illness who took Sertraline according to Japanese Package Insert
Arm/Group | With Past Medical History of Other Illness | Without Past Medical History of Other Illness
Number analyzed (Participants) | 349 | 1808
participants | 57 | 206
Statistical Analysis 1: Comparison: With Past Medical History of Other Illness vs Without Past Medical History of Other Illness; The risk factor tested was "past medical history of other illness". The null hypothesis is there is no difference between "with and without past medical history of other illness" in the participants of responders; Test type: Superiority or Other; p = 0.010, Chi-squared — not adjusted, p=0.050

7. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Average Daily Dose
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether average daily dose is significant risk factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- <25mg: Participants who took less than 25mg of Sertraline a day on average according to Japanese Package Insert
- >=25mg, <50mg: Participants who took more than 25mg and less than 50mg of Sertraline a day on average according to Japanese Package Insert
- >=50mg, <75mg: Participants who took more than 50mg and less than 75mg of Sertraline a day on average according to Japanese Package Insert
- >=75mg, <100mg: Participants who took more than 75mg and less than 100mg of Sertraline a day on average according to Japanese Package Insert
- >=100mg: Participants who took more than 100mg of Sertraline a day on average according to Japanese Package Insert
Arm/Group | <25mg | >=25mg, <50mg | >=50mg, <75mg | >=75mg, <100mg | >=100mg
Number analyzed (Participants) | 28 | 1049 | 590 | 455 | 35
participants | 6 | 175 | 61 | 20 | 1
Statistical Analysis 1: Comparison: <25mg vs >=25mg, <50mg vs >=50mg, <75mg vs >=75mg, <100mg vs >=100mg; The risk factor tested was "average daily dose". The null hypothesis is there is no difference of five types of average daily dose in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

8. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Suicidal Ideation (Including Suicide Attempt)
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without suicidal ideation (including suicide attempt) is significant risk factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Suicidal Ideation (Including Suicide Attempt): Participants with suicidal ideation (including suicide attempt) who took Sertraline according to Japanese Package Insert
- Without Suicidal Ideation (Including Suicide Attempt): Participants without suicidal ideation (including suicide attempt) who took Sertraline according to Japanese Package Insert
Arm/Group | With Suicidal Ideation (Including Suicide Attempt) | Without Suicidal Ideation (Including Suicide Attempt)
Number analyzed (Participants) | 469 | 1608
participants | 73 | 182
Statistical Analysis 1: Comparison: With Suicidal Ideation (Including Suicide Attempt) vs Without Suicidal Ideation (Including Suicide Attempt); The risk factor tested was "suicidal ideation (including suicide attempt)". The null hypothesis is there is no difference between "with and without suicidal ideation(including suicide attempt)" in the participants of responders; Test type: Superiority or Other; p = 0.014, Chi-squared — not adjusted, p=0.050

9. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: 15 Years and Higher of Age or Not
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether 15 years and higher of age or not is significant risk factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- 15 Years and Higher: Participants 15 years and higher of age who took Sertraline according to Japanese Package Insert
- Under 15 Years: Participants under 15 years of age who took Sertraline according to Japanese Package Insert
Arm/Group | 15 Years and Higher | Under 15 Years
Number analyzed (Participants) | 2153 | 4
participants | 261 | 2
Statistical Analysis 1: Comparison: 15 Years and Higher vs Under 15 Years; The risk factor tested was "15 years and higher of age or not". The null hypothesis is there is no difference between "15 years and higher of age or not" in the participants of responders; Test type: Superiority or Other; p = 0.021, Chi-squared — not adjusted, p=0.050

10. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Target Disease Severity
Description: Number of participants with responders of Sertraline to determine whether target disease severity is significant factor
Time Frame: Baseline up to 16 weeks
Population: The efficacy analysis population consists of the evaluable cases in accordance with the analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Groups:
- Mild: Participants whose target disease are mild and who took Sertraline according to Japanese Package Insert
- Moderate: Participants whose target disease are moderate and who took Sertraline according to Japanese Package Insert
- Severe: Participants whose target disease are severe and who took Sertraline according to Japanese Package Insert
Arm/Group | Mild | Moderate | Severe
Number analyzed (Participants) | 478 | 1160 | 127
participants | 416 | 1000 | 93
Statistical Analysis 1: Comparison: Mild vs Moderate vs Severe; The factor tested was "target disease severity". The null hypothesis is there is no difference between "three grade of target disease severity" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

11. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: History of Treatment Prior to Administration of Sertraline Hydrochloride
Description: Number of participants with responders of Sertraline to determine whether with or without history of treatment prior to administration of Sertraline hydrochloride is significant factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Groups:
- With History of Treatment Prior to Sertraline: Participants with history of treatment prior to administration of Sertraline who took Sertraline according to Japanese Package Insert
- Without History of Treatment Prior to Sertraline: Participants without history of treatment prior to administration of Sertraline who took Sertraline according to Japanese Package Insert
Arm/Group | With History of Treatment Prior to Sertraline | Without History of Treatment Prior to Sertraline
Number analyzed (Participants) | 489 | 1202
participants | 398 | 1046
Statistical Analysis 1: Comparison: With History of Treatment Prior to Sertraline vs Without History of Treatment Prior to Sertraline; The factor tested was "history of treatment prior to Sertralin". The null hypothesis is there is no difference between "with and without history of treatment prior to Sertralin" in the participants of responders; Test type: Superiority or Other; p = 0.003, Chi-squared — not adjusted, p=0.050

12. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Outpatient/Inpatient
Description: Number of participants with responders of Sertraline to determine whether outpatient or inpatient is significant factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Groups:
- Inpatient: Participants as inpatients who took Sertraline according to Japanese Package Insert
- Outpatient: Participants as outpatients who took Sertraline according to Japanese Package Insert
Arm/Group | Inpatient | Outpatient
Number analyzed (Participants) | 127 | 1638
participants | 99 | 1410
Statistical Analysis 1: Comparison: Inpatient vs Outpatient; The factor tested was "outpatient or inpatient". The null hypothesis is there is no difference between "outpatient or inpatient" in the participants of responders; Test type: Superiority or Other; p = 0.012, Chi-squared — not adjusted, p=0.050

13. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Complication ;Complications is the Patient's Current Experiences With Illnesses, Operations, Injuries and Treatments.
Description: Number of participants with responders of Sertraline to determine whether with or without complication is significant factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | With Complications | Without Complications
Number analyzed (Participants) | 637 | 1128
participants | 528 | 981
Statistical Analysis 1: Comparison: With Complications vs Without Complications; The factor tested was "complications". The null hypothesis is there is no difference between "with or without complications" in the participants of responders; Test type: Superiority or Other; p = 0.019, Chi-squared — not adjusted, p=0.050

14. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: 15 Years and Higher of Age or Not
Description: Number of participants with responders of Sertraline to determine whether 15 years and higher of age or not is significant factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | 15 Years and Higher | Under 15 Years
Number analyzed (Participants) | 1762 | 3
participants | 1508 | 1
Statistical Analysis 1: Comparison: 15 Years and Higher vs Under 15 Years; The factor tested was "15 years and higher of age or not". The null hypothesis is there is no difference between "15 years and higher of age or not" in the participants of responders; Test type: Superiority or Other; p = 0.010, Chi-squared — not adjusted, p=0.050

15. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Age
Description: Number of participants with responders of Sertraline to determine whether age is significant factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Groups:
- Under 18 Years of Age: Participants under 18 years of age who took Sertraline according to Japanese Package Insert
- 18-44 Years of Age: Participants from 18 to 44 years of age who took Sertraline according to Japanese Package Insert
- 45-64 Years of Age: Participants from 45 to 64 years of age who took Sertraline according to Japanese Package Insert
- Over 65 Years of Age: Participants over 65 years of age who took Sertraline according to Japanese Package Insert
Arm/Group | Under 18 Years of Age | 18-44 Years of Age | 45-64 Years of Age | Over 65 Years of Age
Number analyzed (Participants) | 34 | 955 | 487 | 289
participants | 23 | 829 | 412 | 245
Statistical Analysis 1: Comparison: Under 18 Years of Age vs 18-44 Years of Age vs 45-64 Years of Age vs Over 65 Years of Age; The factor tested was "age". The null hypothesis is there is no difference between "four groups of age" in the participants of responders; Test type: Superiority or Other; p = 0.015, Chi-squared — not adjusted, p=0.050

16. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Suicidal Ideation (Including Suicide Attempt)
Description: Number of participants with responders of Sertraline to determine whether with or without suicidal ideation (including suicide attempt) is significant factor
Time Frame: Baseline up to 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | With Suicidal Ideation (Including Suicide Attempt) | Without Suicidal Ideation (Including Suicide Attempt)
Number analyzed (Participants) | 397 | 1303
participants | 319 | 1136
Statistical Analysis 1: Comparison: With Suicidal Ideation (Including Suicide Attempt) vs Without Suicidal Ideation (Including Suicide Attempt); The factor tested was "suicidal ideation (including suicide attempt)". The null hypothesis is there is no difference between "with or without suicidal ideation (including suicide attempt)" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Sertraline: Participants taking Sertraline according to Japanese Package Insert. All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Arm/Group | Sertraline
Serious Adverse Events (participants affected / at risk) | 9/2157
Other Adverse Events (participants affected / at risk) | 263/2157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=2157)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 1 (1)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=2157)
Nausea (Gastrointestinal disorders) | 87 (87)
Diarrhoea (Gastrointestinal disorders) | 27 (27)
Somnolence (Nervous system disorders) | 23 (23)
Constipation (Gastrointestinal disorders) | 21 (21)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11)
Mania (Psychiatric disorders) | 10 (10)
Malaise (General disorders) | 9 (9)
Headache (Nervous system disorders) | 8 (8)
Dizziness (Nervous system disorders) | 8 (8)
Irritability (General disorders) | 8 (8)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7)
Palpitations (Cardiac disorders) | 6 (6)
Tremor (Nervous system disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Feeling abnormal (General disorders) | 4 (4)
Extrapyramidal disorder (Nervous system disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 3 (3)
Ejaculation delayed (Reproductive system and breast disorders) | 3 (3)
Chest discomfort (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Akathisia (Nervous system disorders) | 2 (2)
Serotonin syndrome (Nervous system disorders) | 2 (2)
Sedation (Nervous system disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Thirst (General disorders) | 2 (2)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Activation syndrome (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Euphoric mood (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Withdrawal syndrome (Psychiatric disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Dysstasia (Nervous system disorders) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.